CLINICAL TRIAL: NCT06079736
Title: A Phase 2, Open-Label, Multiple Ascending Dose Study of PGN-EDO51 With a Long-Term Extension in Participants With Duchenne Muscular Dystrophy Amenable to Exon 51-Skipping Treatment (CONNECT1-EDO51)
Brief Title: A Study Of PGN-EDO51 In Participants With Duchenne Muscular Dystrophy Amenable To Exon 51-Skipping Treatment
Acronym: CONNECT1-EDO51
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PGN-EDO51 development terminated by Sponsor
Sponsor: PepGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PGN-EDO51-102
Record Dates: First submitted 2023-09-29; First posted 2023-10-12 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Enhanced Delivery Oligonucleotide; Peptide-conjugated phosphorodiamidate; Morpholino oligomer; Oligonucleotide; Exon 51; Next-generation oligonucleotide; Cell-penetrating peptide; Muscular Dystrophies; Neuromuscular Disease; Dystrophin production; Splice correcting oligonucleotide; Endosomal Escape; Delivery to the cell nucleus; Antisense oligonucleotide; phosphorodiamidate morpholino oligomer (PPMO)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PGN-EDO51 at Dose Level 1 every 4 weeks (Experimental)
  Interventions: Drug: PGN-EDO51
- PGN-EDO51 at Dose Level 2 every 4 weeks (Experimental)
  Interventions: Drug: PGN-EDO51

INTERVENTIONS:
Drug: PGN-EDO51 — IV infusion

SUMMARY:
The study consists of 3 periods: A Screening Period (up to 45 days), a Multiple Ascending Dose (MAD) Period (16 weeks), and a Long-Term Extension (LTE) Period (108 weeks).

The primary purpose of the MAD period is to evaluate the safety and tolerability of multiple ascending intravenous (IV) doses of PGN-EDO51 administered to participants with Duchenne Muscular Dystrophy (DMD). The primary purpose of the LTE period is to evaluate the long-term safety and tolerability of PGN-EDO51 in participants who have completed the MAD period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DMD able to be corrected by skipping Exon 51
* Body weight at least 18kg at Screening
* Performance of Upper Limb (PUL) 2.0 entry score of at least 4 at Screening (assessing upper limb function in ambulant and non-ambulant individuals with DMD)

Exclusion Criteria:

* Known history or presence of any clinically significant conditions that may interfere with study safety assessments
* Treatment with any gene replacement therapy for the treatment of DMD at any time
* Current or recent systemic infection within 2 weeks prior to Screening or infection requiring IV antibiotics within 4 weeks prior to Screening
* Recent surgery requiring anesthesia within 3 months prior to Screening or expected surgery requiring general anesthesia during the study

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events (safety and tolerability of PGN-EDO51 in MAD period) | Baseline to Week 16
  Adverse events and serious adverse events
Adverse events and serious adverse events (long-term safety and tolerability of PGN-EDO51 in LTE period) | Baseline to Week 108
  Adverse events and serious adverse events

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 12
  Maximum observed plasma concentration of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 12
  Time to maximum observed plasma concentration of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 12
  Apparent terminal half-life of PGN-EDO51
Plasma pharmacokinetic (PK) parameters (MAD period) | Baseline to Week 12
  Area under the curve for concentration time of PGN-EDO51
PK Plasma levels (LTE period) | Baseline to Week 104
  PK sampling for PGN-EDO51 and PGN-PMO51 plasma levels
Skeletal muscle concentration of PGN-EDO51 (MAD period) | Baseline to Week 16
  Change from baseline in skeletal muscle concentration of PGN-EDO51 after multiple doses
Dystrophin Levels (MAD period) | Baseline to Week 16
  Change from baseline in dystrophin levels measured after multiple doses

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - CHU de Québec, Québec, Quebec